CLINICAL TRIAL: NCT00131885
Title: Effects of St. John's Wort on Levonorgestrel
Brief Title: Effects of St. John's Wort on the Oral Contraceptive Hormone Levonorgestrel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Patricia Murphy, Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13430; R21AT002297 (NIH)
Record Dates: First submitted 2005-08-17; First posted 2005-08-19 (Estimated); Results first posted 2010-06-09 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Contraception
Keywords: Menstruation; Complementary Therapies; Pharmacokinetics; Hypericum; St. John's wort; Levonorgestrel; Women
MeSH Terms: interventions — Hypericum extract LI 160; Levonorgestrel

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Levonorgestrel 1.5 with Placebo Herb (Placebo Comparator): This group had baseline pharmacokinetic studies after an oral dose of levonorgestrel (LNG) 1.5 mg, then took a placebo herb daily for 4-6 weeks, during which time pharmacokinetic studies were repeated after an oral dose of LNG 1.5 mg
  Interventions: Dietary Supplement: Placebo Control (Placebo Herb); Drug: Levonorgestrel
- Levonorgestrel 1.5 with SJW 900 mg (Active Comparator): This group had baseline pharmacokinetic studies after an oral dose of levonorgestrel (LNG) 1.5 mg, then took St. John's Wort (SJW) 900 mg a Day orally for 4-6 weeks, during which time pharmacokinetic studies were repeated after an oral dose of LNG 1.5 mg
  Interventions: Dietary Supplement: St. John's Wort; Drug: Levonorgestrel
- Levonorgestrel 2.25 with SJW 900 mg (Active Comparator): This group had baseline pharmacokinetic studies after an oral dose of levonorgestrel (LNG) 1.5 mg, then took a St. Johns's Wort 300 mg capsules three times daily for 4-6 weeks, during which time pharmacokinetic studies were repeated after an oral dose of LNG 2.25 mg
  Interventions: Dietary Supplement: St. John's Wort; Drug: Levonorgestrel
- Levonorgestrel 1.5 with SJW 1500 mg (Active Comparator): This group had baseline pharmacokinetic studies after an oral dose of levonorgestrel (LNG) 1.5 mg, then took a St. Johns's Wort 300 mg capsules five times daily for 4-6 weeks, during which time pharmacokinetic studies were repeated after an oral dose of LNG 1.5 mg
  Interventions: Dietary Supplement: St. John's Wort; Drug: Levonorgestrel

INTERVENTIONS:
Dietary Supplement: Placebo Control (Placebo Herb) — Placebo herb three times daily (ground cellulose) for 4-6 weeks
  Arms: Levonorgestrel 1.5 with Placebo Herb
Dietary Supplement: St. John's Wort — St. John's Wort (Hypericum perforatum) orally or 4-6 weeks
  Arms: Levonorgestrel 1.5 with SJW 1500 mg; Levonorgestrel 1.5 with SJW 900 mg; Levonorgestrel 2.25 with SJW 900 mg
Drug: Levonorgestrel — Levonorgestrel in a single oral dose

SUMMARY:
This study will determine the effects of St. John's wort, a common herbal remedy, on metabolism of the female contraceptive hormone levonorgestrel.

DETAILED DESCRIPTION:
In the last decade, St. John's wort has become one of the most commonly used botanicals. Levonorgestrel is a form of progesterone, a female hormone involved in conception. It can be given as both a pill and an injection and is used for contraception and for the treatment of endometriosis. However, evidence suggests that St. John's wort may reduce the effectiveness of the contraceptive hormone levonorgestrel. This study will determine whether interactions between St. John's wort and levonorgestrel reduce the effectiveness of the hormone. This study will also determine whether a higher dose of levonorgestrel will override the effects of St. John's wort.

All participants will receive a single dose of levonorgestrel between Days 9 and 12 of their first menstrual cycle after entering this study. Blood and urine collection will occur immediately after the levonorgestrel is given and every week until participants' next menstrual cycle to determine the levels of reproductive hormones in participants' bodies.

At the beginning of participants' next menstrual cycle, they will be randomly assigned to one of four groups and receive either St. John's wort or placebo for 6 weeks. Group 1 will receive a placebo; Groups 2 and 3 will receive a standard dose of St. John's wort (900 mg per day); and Group 4 will receive an increased dose of St. John's wort (1500 mg per day). After 6 weeks, Groups 1, 2, and 4 will receive 150 mcg levonorgestrel; and Group 3 will receive 225 mcg levonorgestrel. Blood and urine collection will occur immediately after levonorgestrel is given and every week until participants' next menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 20 and 25
* Regular menstrual cycles for at least 3 months prior to study entry

Exclusion Criteria:

* Current use of foods, herbs, vitamins, over-the-counter supplements, or any medications that could alter pharmacokinetics of other drugs
* Medical contraindications to the use of contraceptives

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2005-08; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A. Murphy, DrPH, Principal Investigator — College of Nursing, University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Murphy PA, Kern SE, Stanczyk FZ, Westhoff CL. Interaction of St. John's Wort with oral contraceptives: effects on the pharmacokinetics of norethindrone and ethinyl estradiol, ovarian activity and breakthrough bleeding. Contraception. 2005 Jun;71(6):402-8. doi: 10.1016/j.contraception.2004.11.004. PMID 15914127

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were recruited via local advertising.
Pre-assignment Details: No enrolled participants were excluded
Groups:
- LNG 1.5 mg Dose, Then Placebo Herb, LNG 1.5 mg: Group 1: one-time oral dose of levonorgestrel 1.5 mg at the first pharmacokinetic study, followed by placebo herb and a one-time oral dose of levonorgestrel 1.5 mg at the second pharmacokinetic study
- LNG 1.5 mg Dose, Then SJW 900 mg Day, LNG 1.5 mg: Group 2: One-time oral dose of levonorgestrel 1.5 mg at the first pharmacokinetic study, followed by St. John's Wort 300 mg orally three times per day, and a one-time oral dose of levonorgestrel 1.5 mg at the second pharmacokinetic study
- LNG 1.5 mg Dose, Then SJW 900 mg Daily, 2.25 mg LNG Dose: Group 3: A one-time oral dose of levonorgestrel 1.5 mg mg at the first pharmacokinetic study, followed by St. John's Wort 300 mg orally three times per day (900 mg total) and a one-time oral dose of levonorgestrel 2.25 mg at the second pharmacokinetic study
- LNG 1.5 mg Dose, Then SJW 1500 ng Day, 1.5 mg LNG: Group 4: A one-time oral dose of levonorgestrel 1.5 mg at the first pharmacokinetic study, then St. John's Wort 300 mg orally five times per day (total 1500 mg daily) and a one-time oral dose of levonorgestrel 1.5 mg at the second pharmacokinetic study
Period: Time 1: First Intervention
Arm/Group | LNG 1.5 mg Dose, Then Placebo Herb, LNG 1.5 mg | LNG 1.5 mg Dose, Then SJW 900 mg Day, LNG 1.5 mg | LNG 1.5 mg Dose, Then SJW 900 mg Daily, 2.25 mg LNG Dose | LNG 1.5 mg Dose, Then SJW 1500 ng Day, 1.5 mg LNG
Started | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Time 2: Second Intervention
Arm/Group | LNG 1.5 mg Dose, Then Placebo Herb, LNG 1.5 mg | LNG 1.5 mg Dose, Then SJW 900 mg Day, LNG 1.5 mg | LNG 1.5 mg Dose, Then SJW 900 mg Daily, 2.25 mg LNG Dose | LNG 1.5 mg Dose, Then SJW 1500 ng Day, 1.5 mg LNG
Started | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LNG 1.5 mg Dose, Then Placebo Herb, LNG 1.5 mg | LNG 1.5 mg Dose, Then SJW 900 mg Day, LNG 1.5 mg | LNG 1.5 mg Dose, Then SJW 900 mg Daily, 2.25 mg LNG Dose | LNG 1.5 mg Dose, Then SJW 1500 ng Day, 1.5 mg LNG | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 9 | 9 | 36
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.1 (3.6) | 22.4 (3.1) | 23 (3.5) | 22.9 (3.4) | 22.9 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 9 | 9 | 36
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 9 | 9 | 36

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Versus Time Curve for 0 to 24 Hours After Drug Administration, Done Between Days 9 and 12 of the Menstrual Cycle at Time 1 (Before) and Time 2 (During Treatment With St. John's Wort or Placebo)
Description: Pharmacokinetic studies were done between Days 9-12 of the menstrual cycle at Time 1 (baseline, before any treatment with herb or placebo), and at Time 2 (intervention, after treatment with herb or placebo). Serum samples drawn at 0, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16, and 24 hours, following oral administration of a dose of levonorgestrel.
  Treatment between the two time periods was with St. John's Wort or placebo herb, beginning after the Time 1 (baseline) and continued for 5 weeks until Time 2.
  Estimates of levonorgestrel clearance were made using a two stage non-compartmental approach to determine individual and group parameters.
Time Frame: Area Under the Concentration versus Time curve for 0 to 24 hours after drug administration, between Days 9 and 12 of the menstrual cycle, done at Time 1 and at Time 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | LNG 1.5 mg Dose, Then Placebo Herb, LNG 1.5 mg | LNG 1.5 mg Dose, Then SJW 900 mg Day, LNG 1.5 mg | LNG 1.5 mg Dose, Then SJW 900 mg Daily, 2.25 mg LNG Dose | LNG 1.5 mg Dose, Then SJW 1500 ng Day, 1.5 mg LNG
Number analyzed (Participants) | 9 | 9 | 9 | 9
ng*hr/mL
  AUC 0-24 hours after drug administration Time 1 | 586.3 (530.6) | 379.4 (201.3) | 339.4 (201.2) | 253.3 (114.4)
  AUC 0-24 hours after drug administration Time 2 | 478.2 (374.0) | 317.4 (171.6) | 439.4 (320.1) | 210.1 (100.4)

2. Primary Outcome: Number of Participants With Progesterone Levels Above 3.0 ng/ml at Time 1 (Baseline) and Time 2 (After Intervention With St John's Wort or Placebo).
Description: Serum progesterone levels were drawn at the time of dosing with levonorgestrel and then at weekly intervals until menses occurred. This was done at Time 1 (baseline), and again at Time 2 (after 5 weeks of dosing with St. John's Wort or placebo).
  Possible ovulation was defined as a serum progesterone >3ng/ml within 2 weeks of Days 9-12 of the menstrual cycle.
Time Frame: Progesterone levels drawn at weekly intervals after dosing with levonorgestrel between Days 9 and 12 of the menstrual cycle, at each time point until menses
Measure: Number; unit: Participants
Arm/Group | LNG 1.5 mg Dose, Then Placebo Herb, LNG 1.5 mg | LNG 1.5 mg Dose, Then SJW 900 mg Day, LNG 1.5 mg | LNG 1.5 mg Dose, Then SJW 900 mg Daily, 2.25 mg LNG Dose | LNG 1.5 mg Dose, Then SJW 1500 ng Day, 1.5 mg LNG
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  Ovulation (Progesterone Levels > 3.0 ng/ml) Time 1 | 3 | 1 | 1 | 3
  Ovulation (Progesterone Levels >3.0 ng/ml) Time 2 | 3 | 2 | 2 | 2

3. Secondary Outcome: Mean Levels of Follicle-stimulating Hormone Drawn at Weekly Intervals Until Next Menses
Description: Descriptive reporting of secondary outcomes of reproductive hormone levels (including FSH, E2, LH).
  Pharmacokinetic studies were done between Days 9-12 of the menstrual cycle at Time 1 (baseline, before any treatment with herb or placebo), and at Time 2 (intervention, after treatment with herb or placebo).
  Weekly means are reported for both time periods at week 0 (day of pharmacokinetic study), week 1 (one week after pharmacokinetic study) and week 2 (2 weeks after pharmacokinetic study).
Time Frame: Time Frame: Time 1 (pre-intervention baseline) and Time 2 (following a 6 week intervention)
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | LNG 1.5 mg Dose, Then Placebo Herb, LNG 1.5 mg | LNG 1.5 mg Dose, Then SJW 900 mg Day, LNG 1.5 mg | LNG 1.5 mg Dose, Then SJW 900 mg Daily, 2.25 mg LNG Dose | LNG 1.5 mg Dose, Then SJW 1500 ng Day, 1.5 mg LNG
Number analyzed (Participants) | 9 | 9 | 9 | 9
IU/mL
  FSH, IU/mL, Time 1, week 0 | 14.9 (5.7) | 14.0 (4.8) | 15.8 (8.0) | 13.9 (4.3)
  FSH, IU/mL, Time 1, week 1 | 14.5 (5.0) | 14.7 (4.8) | 13.9 (5.2) | 13.6 (4.4)
  FSH, IU/mL, Time 1, week 2 | 13.8 (4.2) | 13.4 (4.3) | 20.4 (12.0) | 15.4 (9.9)
  FSH, IU/mL, Time 2, week 0 | 12.9 (3.5) | 13.0 (3.6) | 17.5 (10.1) | 14.7 (4.1)
  FSH, IU/mL, Time 2, week 1 | 11.8 (3.0) | 15.9 (5.0) | 17.7 (8.8) | 13.8 (4.5)
  FSH, IU/mL, Time 2, week 2 | 11.3 (4.4) | 14.1 (4.5) | 14.8 (4.7) | 16.8 (10.1)

4. Primary Outcome: Clearance (L/hr) of Levonorgestrel Over 24 Hours for Each Dosage Group and Each Study Session.
Description: Average and standard deviation for Clearance (L/hr) of Levonorgestrel study for each dosage group and each study session.
Time Frame: Time Frame: Time 1 (pre-intervention baseline) and Time 2 (following a 6 week intervention)
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | LNG 1.5 mg Dose, Then Placebo Herb, LNG 1.5 mg | LNG 1.5 mg Dose, Then SJW 900 mg Day, LNG 1.5 mg | LNG 1.5 mg Dose, Then SJW 900 mg Daily, 2.25 mg LNG Dose | LNG 1.5 mg Dose, Then SJW 1500 ng Day, 1.5 mg LNG
Number analyzed (Participants) | 9 | 9 | 9 | 9
L/hr
  Clearance (L/hr) Time 1 | 4.06 (2.60) | 4.93 (2.19) | 6.39 (4.23) | 6.85 (2.51)
  Clearance L/hr Time 2 | 4.64 (2.44) | 5.63 (2.08) | 7.68 (4.97) | 8.92 (4.60)

5. Secondary Outcome: Mean Levels of Estradiol-17b (E2) Drawn at Weekly Intervals Until Next Menses
Description: as for outcome 3
Time Frame: Time Frame: Time 1 (pre-intervention baseline) and Time 2 (following a 6 week intervention)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | LNG 1.5 mg Dose, Then Placebo Herb, LNG 1.5 mg | LNG 1.5 mg Dose, Then SJW 900 mg Day, LNG 1.5 mg | LNG 1.5 mg Dose, Then SJW 900 mg Daily, 2.25 mg LNG Dose | LNG 1.5 mg Dose, Then SJW 1500 ng Day, 1.5 mg LNG
Number analyzed (Participants) | 9 | 9 | 9 | 9
pg/mL
  Estradiol, pg/mL, Time 1, week 0 | 133.3 (64.3) | 137.2 (76.9) | 131.1 (75.0) | 103.5 (52.2)
  Estradiol, pg/mL, Time 1, week 1 | 142.2 (90.0) | 154.7 (117.1) | 138.4 (77.7) | 290.6 (34.8)
  Estradiol, pg/mL,Time 1, week 2 | 132.4 (103.9) | 107.9 (39.3) | 132.6 (73.3) | 230.4 (34.2)
  Estradiol, pg/mL,Time 2, week 0 | 134.2 (73.9) | 102.0 (44.2) | 119.3 (77.9) | 123.4 (60.2)
  Estradiol, pg/mL,Time 2, week 1 | 210.7 (227.1) | 121.6 (57.5) | 113.9 (71.1) | 118.0 (86.3)
  Estradiol, pg/mL,Time 2, week 2 | 146.3 (80.5) | 192.0 (101.2) | 102.9 (75.1) | 108.7 (47.6)

6. Secondary Outcome: Mean Levels of Luteinizing Hormone, Drawn at Weekly Intervals Until Next Menses
Description: as for outcome 3
Time Frame: Time Frame: Time 1 (pre-intervention baseline) and Time 2 (following a 6 week intervention)
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | LNG 1.5 mg Dose, Then Placebo Herb, LNG 1.5 mg | LNG 1.5 mg Dose, Then SJW 900 mg Day, LNG 1.5 mg | LNG 1.5 mg Dose, Then SJW 900 mg Daily, 2.25 mg LNG Dose | LNG 1.5 mg Dose, Then SJW 1500 ng Day, 1.5 mg LNG
Number analyzed (Participants) | 9 | 9 | 9 | 9
IU/mL
  LH, IU/L, Time 1, week 0 | 24.7 (10.1) | 20.9 (10.4) | 26.4 (15.7) | 25.3 (15.7)
  LH, IU/L, Time 1, week 1 | 35.1 (16.1) | 30.2 (21.8) | 24.6 (16.3) | 25.3 (15.7)
  LH, IU/L, Time 1, week 2 | 36.2 (20.1) | 23.1 (14.7) | 25.6 (22.1) | 23.2 (18.4)
  LH IU/L, Time 2, week 0 | 33.2 (16.5) | 28.4 (14.9) | 31.9 (27.5) | 46.3 (25.8)
  LH, IU/L, Time 2, week 1 | 30.1 (20.0) | 27.5 (17.9) | 40.0 (46.5) | 28.8 (11.4)
  LH, IU/L, Time 2, week 2 | 29.1 (22.5) | 27.7 (19.1) | 27.7 (19.1) | 39.1 (18.0)

ADVERSE EVENTS:
Arm/Group | LNG 1.5 mg Dose, Then Placebo Herb, LNG 1.5 mg | LNG 1.5 mg Dose, Then SJW 900 mg Day, LNG 1.5 mg | LNG 1.5 mg Dose, Then SJW 900 mg Daily, 2.25 mg LNG Dose | LNG 1.5 mg Dose, Then SJW 1500 ng Day, 1.5 mg LNG
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No